CLINICAL TRIAL: NCT06467877
Title: Retrospective Analysis of Causes, Clinical Presentation and Treatment in Patients With Hypercalcaemia in the Emergency Department of a Tertiary German Hospital
Brief Title: Causes, Characteristics and Treatment of Hypercalcemia in the Emergency Room of a German Hospital
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, Prof. Dr. med., University of Cologne
Other Study IDs: V1.0-13.05.2024
Record Dates: First submitted 2024-06-14; First posted 2024-06-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Hypercalcemia
Keywords: hypercalcemia; calcium; emergency room; mortality
MeSH Terms: conditions — Hypercalcemia; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective Chart Review: Group includes patient with hypercalcemia ≥2.65 mmol/l, who reported to the emergency room of a tertiary hospital

SUMMARY:
Patients with hypercalcemia were identified in the patient population of a German emergency department during a 11 year time period and studied regarding reproducibility of elevated calcium values, causes of hypercalcemia, symptoms. acute renal injury, mortality and treatment response.

DETAILED DESCRIPTION:
Patients, who presented to the emergency department of a tertiary German hospital with a total calcium of ≥2.65 mmol/l between January 2010 and March 2021, was retrospectively studied. From the electronic patient records we analyzed if the elevated calcium values were reproducible in follow-up measurements, identified the cause of hypercalcemia, listed the symptoms, investigated a correlation between calcium and creatinine values to study acute renal injury directly due to hypercalcemia, calculated the mortality rate stratified by the calcium value on presentation and studied the treatment response regarding lowering calcium values by different treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Total calcium ≥ 2.65 mmol/l
* Female and male

Exclusion Criteria:

* Age < 18 years
* Total calcium < 2.65 mmol/

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients reporting to the Emergency Room of the University Hospital Cologne and recieved a determination of the total calcium level
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of total calcium values | 5 days after enrollment
  Overview of total calcium values within 5 days

SECONDARY OUTCOMES:
Reproducibility of elevated calcium values | 5 days after enrollment
  Determination of cause of hypercalcemia, of symptoms, of treatment response. In dependence of hospital stay, kann be determined later than 5 days after enrollment
Correlation creatinine calcium | 5 days after enrollment
  Determination of correlation between calcium and creatinine.
Mortality | 5 days after enrollment
  occurence of death within of 5 days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Principal Investigator — University Hospital of Cologne
Locations (1):
- Department II of Internal Medicine,University of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No